CLINICAL TRIAL: NCT03407508
Title: Control of Diabetes and Periodontitis Through a New Anti-inflammatory Nordic Diet
Brief Title: Diet, Diabetes and Periodontitis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kristianstad University (Other)
Responsible Party: Principal Investigator, Cecilia Widen, Principal Investigator, Kristianstad University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2017/540
Record Dates: First submitted 2018-01-03; First posted 2018-01-23 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Diabetes Mellitus; Gingivitis
MeSH Terms: conditions — Diabetes Mellitus; Gingivitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (Placebo Comparator): No dietary changes.
  Interventions: Dietary Supplement: Comparison of Diets
- Comparison of Diets (Placebo Comparator): Okinawan-based Nordic Diet or Control Diet.
  Interventions: Dietary Supplement: Comparison of Diets

INTERVENTIONS:
Dietary Supplement: Comparison of Diets — Okinawan-based Nordic Diet and Control Diet

SUMMARY:
There is a significant and growing interest in nutrition and health in the general population and there is also, paradoxically, an increasing problem with obesity and general debilitating conditions of affluence, such as type 2 diabetes mellitus. Igelösa Life Science AB has developed a modified Okinawan-based Nordic Diet (OBND) diet based on evidence primarily from the diet of the long-lived and healthy Okinawa population. The diet includes fish and whole grains, with a high level of vegetables, but is low in fat. In 2016, a clinical nutrition study was carried out at Kristianstad University with the intention to determine if the OBND resulted in reductions/changes in clinical and medical markers of importance for treatment of diabetes mellitus and gingivitis/periodontitis. The diet had a positive impact on the clinical progress of otherwise debilitating conditions such as diabetes and the health benefits on clinical parameters was extremely rapid, that is, within two weeks. Not only did the patients with type 2 diabetes receive the OBND, their partners were also offered the same option. This is a key innovation and the participants stated that it was a great support, which facilitated adherence and promotes the long-term impact on health. Ingrained habits such as poor diet, can only be defeated by a concerted team effort and our work to date provides a glimpse of the potential benefits to Sweden and the rest of the developed world through this shared approach.

Initial studies have shown promising effects of the OBND on both diabetes and periodontal conditions. The objective of this study is to compare the OBND to the current recommended standard diet. Assuming the study provides positive evidence of health impact due to improved food quality, it will also be seen that the production and delivery of such 'healthy-living' meals will be of commercial interest for industry. The mission is to offer an evidence-based natural food alternative that both prevents disease and improves the health status of individuals with diabetes. The long-term goal is to design efficient and effective products that will protect against diabetes and other chronic diseases. The combination of scientific credibility and commercial interests may be a key factor to transfer the new knowledge about healthy dieting into actual improvements in public health.

DETAILED DESCRIPTION:
The project has one main goal: to perform a clinical trial to compare the OBND with standard of care diet. The outcome of the clinical trial will be analyzed in the areas: medicine/odontology, sensory science, nursing, public health and health economics.

Study objectives:

* To assess if the consumption of the designated diet results in added medical/dental health outcome for the OBND in comparison to standard of care diet. The study is a randomized case control clinical trial.
* To perform cost-effectiveness analyses comparing costs and health benefits for the test and control diets with focus on individuals with type 2 diabetes mellitus and otherwise healthy individuals living in close relationship to those with diabetes.
* To assess consumer acceptance of the diet: (I) acceptance of the diets (questionnaire, focus groups and food diary), (II) acceptability of the diet in relation to taste of the diet, and the prospect of adopting the diet in everyday life, and (III) sensory analysis of identical dishes prepared according to the OBND and the standard of care diet.

Study design The study design is a randomized double-blinded clinical trial with four subgroups including 20 individuals per study group.

Test Group A: OBND, individuals diagnosed with type 2 diabetes (T2D) with a need for insulin intake

Test Group B: OBND, relatives who do not have T2D

Control Group C: Standard of care diet, individuals diagnosed with T2D with a need for insulin intake

Control Group D: Standard of care diet, relatives who do not have T2D

Based on the above reported studies and available data on blood sugar and lipid values, the investigators have identified that 18 individuals in each group will provide adequate statistical power (alpha=0.05, beta=0.85). While lost to follow up occurs, the investigators will enroll 20 individuals in each group. Thus, a total of 80 study individuals (test and control) will be enrolled. Data analyses will be performed according to per protocol as well as per intent to treat. Clinical examination procedures in medicine and dentistry will follow principles of good clinical practice. Study group assignment will be based on a randomization using the SPSS statistics package. A pre-baseline examination will be performed to ensure that all study individuals fulfill study requirements. The investigators will monitor that study individuals are compliant to protocol.

Study time schedule The study design includes a pre-baseline study examination two weeks before study start to ensure that study individuals meet the criteria for study participation and to control for Hawthorne effects. Study individuals will be enrolled in groups of 8 to 10 individuals and re-examined at baseline. The primary study endpoint is the third examination will be performed 4 weeks after baseline examination. A follow-up examination will occur after 6 months (plus/minus 14 days). All study enrollments will be completed within one month. Study individuals will receive phone calls during the study period to encourage compliance and respond to specific questions.

ELIGIBILITY:
Inclusion Criteria:

* minimum 20 teeth
* HbA1c = 60-80 mmol/mol (diabetics), HbA1c < 42 mmol/mol (control)
* be able to receive food delivery monday, wednesday, friday
* Scandinavian background

Exclusion Criteria:

* use of tobacco products
* pregnancy
* lactose, celiac- or garlic intolerance
* blood pressure ≥ 180 mm Hg
* have visited dental clinic within one month Before study start or currently are undergoing dental/dental hygienist treatment
* have rheumatoid arthritis
* for Medical reasons need treatment with antibiotics or who has been treated with antiobiotics within one month before study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-10-17 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
HbA1c | Baseline, 2, 4, and 26 weeks
  Changes in levels of HbA1c (mmol/mol) in serum before and after study procedures

SECONDARY OUTCOMES:
Pro-inflammatory cytokines | Baseline, 2, 4, and 26 weeks
  Change in levels of pro-inflammatory cytokines (pg/ml) in serum and gingival fluid in relation to gingival bleeding, before and after study procedures
Gingivitis | Baseline, 2, 4, and 26 weeks
  Changes in the extent of gingivitis, as determined by the severity of gingival bleeding (%), before and after the study procedures

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kristianstad, Kristianstad, Skåne County, Sweden